CLINICAL TRIAL: NCT01572350
Title: Randomized Multicenter Clinical Trial of Three Parallel Groups to Estimate the Safety and Efficacy of Triamcinolone Acetonide Combined With Laser, Bevacizumab Combined With Laser Versus Laser Alone for the Treatment of Diffuse Non-tractional Diabetic Macular Edema.
Brief Title: Safety and Efficacy of Triamcinolone Acetonide Combined With Laser, Bevacizumab Combined With Laser Versus Laser Alone for the Treatment of Diffuse Non-tractional Diabetic Macular Edema
Acronym: ALBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALBA09
Record Dates: First submitted 2011-04-07; First posted 2012-04-06 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Triamcinolone Acetonide; Triamcinolone; Bevacizumab

ARMS (3):
- Grid laser (Active Comparator): It's a reference standard as the treatment which is currently accepted for NTDDME
  Interventions: Other: Grid laser
- Triamcinolone 4 mg (Experimental)
  Interventions: Drug: Triamcinolone Acetonide
- Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Other: Grid laser — Grid laser therapy acts as the standard to refer to as it is the treatment which is currently accepted by EMDDNT.
  Arms: Grid laser
Drug: Triamcinolone Acetonide — Triamcinolone 4 mg followed by modified grid laser therapy after 3-4 weeks
  Other Names: Triesence
  Arms: Triamcinolone 4 mg
Drug: Bevacizumab — Bevacizumab (1.25 mg initially, weeks 6 and 12) followed by modified grid laser therapy after3-4 weeks
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
This clinical trial is designed to investigate differences in terms of efficacy (mean change in best corrected visual acuity obtained after 12 months of treatment) and safety, of 3 therapeutic estrategies for non-tractional macular edema in diabetic patients: a) laser alone; b) laser plus tiramcinolon; and c) laser plus bevacizumab.

ELIGIBILITY:
To be eligible, the following inclusion criteria must be met:

1. Age ≥18 years from both sexes. Women of childbearing age should use adequate contraception methods and submit a negative pregnancy test.
2. Diagnosis of diabetes mellitus type 1 or type 2 (documented by ADA or WHO guidelines) and serum HbA1c <11% at the time of randomization (determinations done in the last two months).
3. Patient able to give informed consent.
4. Eye with clear media, pupil dilation and patient able to cooperate to perform retinography, OCT and fluorescein angiography.
5. Patients with clinically significant diabetic macular edema; the patient must have at least one:

   5.1) retinal thickening within 500 μ from the center or 5.2) hard exudates within 500 μ from the center if associated with adjacent retinal thickening or 5.3) the size of retinal thickening at least 1 area disc, part of which is less than 1 DD of the center.
6. Patients with diffuse diabetic macular edema.
7. Patients with not tractional diabetic macular edema.

A patient is not eligible if any of the following exclusion criteria are present:

1. Women of childbearing age not using adequate contraceptive methods.
2. Pregnancy and lactation. Pregnancy test was performed before starting treatment.
3. Chronic renal failure requiring dialysis or kidney transplantation.
4. Allergy to any of the drugs included in the study.
5. Systemic use of steroids in the last 4 months.
6. Patient intends to change his place of residence within 3 years after recruitment, whenever you go to an area not covered by the study.
7. Blood pressure>180/110. If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.
8. HbA1c> 11% in the current analysis or done in the last 2 months.
9. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hare exudates, nonretinal condition).
10. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.)
11. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more
12. History of prior treatment with intravitreal corticosteroids or intravitreal antiangiogenic.
13. History of peribulbar steroid injection within 6 months prior to randomization.
14. History of focal, grid or panretinal photocoagulation within 4 months prior to randomization.
15. Need of panretinal photocoagulation in the first 4 months of treatment.
16. History of prior pars plana vitrectomy.
17. Major ocular surgery (including cataract extraction, scleral buckle, vitrectomy, etc.) within prior 6 months or anticipated within the next 6 months following randomization.
18. History of YAG capsulotomy performed within 2 months prior to randomization.
19. Intraocular pressure >25mmHg.
20. History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion). A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is <25 mmHg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous.
21. History of cortisone-induced glaucoma that required IOP-lowering treatment.
22. History of prior herpetic ocular infection.
23. Exam evidence of ocular toxoplasmosis.
24. Aphakia.
25. Presence of pseudoexfoliation.
26. Evidence of external ocular infection, including: conjunctivitis, chalazion and blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2010-10 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | 12 months
  To evaluate the effect on best-corrected visual acuity (BCVA) of intravitreal triamcinolone (Triesence ®) or bevacizumab (Avastin ®) in combination with grid laser therapy compared to grid laser therapy alone after 12 months of treatment, in diabetic patients with not tractional diffuse macular edema (NTDDEM)

SECONDARY OUTCOMES:
To assess the safety of intravitreal Triesence (r) | Baseline, 3m, 6m and 12 months
  Type of adverse events, severity and number of Participants with Adverse Events as a Measure of Safety and Tolerability.
To measure average change in mean central macular thickness in each group. | Baseline and 3, 6 and 12 months after the treatment was initiated.
  To measure average change in mean central macular thickness (in microns) obtained by Optical Coherence Tomography (OCT) at each follow-up visits compared to the baseline visit in each of the three groups.
To assess the safety of intravitreal Avastin (r) | Baseline, 3m, 6m and 12 months
  Type of adverse events, severity and number of Participants with Adverse Events as a Measure of Safety and Tolerability
To assess the safety of intravitreal grid photocoagulation | Baseline, 3m, 6m and 12 months
  Type of adverse events, severity and number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Pareja, MD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario Dr Negrín, Las Palmas de Gran Canaria, Spain

REFERENCES:
- [Derived] Pareja-Rios A, de Armas-Ramos E, Aldea-Perona A, Bonaque-Gonzalez S. Alone laser versus bevacizumab plus laser for diffuse diabetic macular edema (ALBA randomized trial). Ther Adv Ophthalmol. 2021 Jan 15;13:2515841420988210. doi: 10.1177/2515841420988210. eCollection 2021 Jan-Dec. PMID 33506177